CLINICAL TRIAL: NCT01583218
Title: (Apex) Multicenter, Randomized, Active-Controlled Efficacy And Safety Study Comparing Extended Duration Betrixaban With Standard Of Care Enoxaparin For The Prevention Of Venous Thromboembolism In Acute Medically Ill Patients
Brief Title: Acute Medically Ill VTE Prevention With Extended Duration Betrixaban Study (The APEX Study)
Acronym: APEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11-019
Record Dates: First submitted 2012-04-16; First posted 2012-04-23 (Estimated); Results first posted 2017-09-20 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Venous Thromboembolism (VTE)
Keywords: Phase III
MeSH Terms: conditions — Venous Thromboembolism | interventions — betrixaban; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Betrixaban (Experimental): Daily oral (PO) betrixaban capsules for 35 to 42 days and subcutaneous (SQ) injections of enoxaparin placebo for 10 ± 4 days
  Interventions: Drug: Betrixaban
- Enoxaparin (Active Comparator): Daily subcutaneous (SQ) injections of enoxaparin for 10 ± 4 days and oral (PO) betrixaban placebo capsules for 35 to 42 days
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Betrixaban — Betrixaban 80 mg PO once daily (QD) for 35 day + 7 days.
  Enoxaparin Placebo: Once daily, 6-14 days
  Arms: Betrixaban
Drug: Enoxaparin — Enoxaparin 40 mg subcutaneous (SC) QD for 10 ± 4 days.
  Betrixaban Placebo: once daily, 35 days
  Arms: Enoxaparin

SUMMARY:
The purpose of this study is to evaluate whether extended prophylaxis with oral betrixaban can prevent blood clots in the leg and lung that sometime occur in patients hospitalized for an acute medical illness and to compare these results with standard of care enoxaparin. The safety of betrixaban will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* men and non-pregnant, non-breastfeeding women
* anticipated to be severely immobilized for at least 24 hours after randomization
* hospitalized with one of the following

  * congestive heart failure
  * acute respiratory failure,
  * acute infection without septic shock,
  * acute rheumatic disorders
  * acute ischemic stroke with lower extremity hemiparesis or hemi paralysis

Exclusion Criteria:

* a condition requiring prolonged anticoagulation or anti-platelets
* active bleeding or at high risk of bleeding
* contraindication to anticoagulant therapy
* general conditions in which subjects are not suitable to participate in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7513 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (371):
- United States (72):
  - Birmingham, Alabama
  - Bakersfield, California
  - Fresno, California
  - La Mesa, California
  - Long Beach, California
  - Los Angeles, California
  - Modesto, California
  - San Diego, California
  - Stanford, California
  - Torrance, California
  - Englewood, Colorado
  - Bay Pines, Florida
  - Clearwater, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Pensacola, Florida
  - Sarasota, Florida
  - Vero Beach, Florida
  - Columbus, Georgia
  - Decatur, Georgia
  - Chicago, Illinois
  - Oak Park, Illinois
  - Carmel, Indiana
  - Davenport, Iowa
  - Windsor Heights, Iowa
  - Topeka, Kansas
  - Hazard, Kentucky
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Detroit, Michigan
  - Grand Blanc, Michigan
  - Royal Oak, Michigan
  - Troy, Michigan
  - Duluth, Minnesota
  - Picayune, Mississippi
  - Kansas City, Missouri
  - St Louis, Missouri
  - Butte, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Reno, Nevada
  - Atlantic City, New Jersey
  - Pomona, New Jersey
  - Somerville, New Jersey
  - Summit, New Jersey
  - Buffalo, New York
  - Manhasset, New York
  - Staten Island, New York
  - Valhalla, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Camp Hill, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Orangeburg, South Carolina
  - Austin, Texas
  - Bellaire, Texas
  - Corsicana, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - McAllen, Texas
  - Mission, Texas
  - San Antonio, Texas
  - Victoria, Texas
  - Colchester, Vermont
  - Charlottesville, Virginia
  - Richmond, Virginia
  - Everett, Washington
  - Huntington, West Virginia
- Argentina (7):
  - Buenos Aires
  - Coronel Suarez, Buenos Aires
  - Corrientes
  - Córdoba
  - El Talar
  - Rosario, Santa Fe
  - San Miguel de Tucumán
- Australia (7):
  - Redcliffe, Queensland
  - Bedford Park, South Australia
  - Nedlands, Western Australia
  - Milton
  - Parkville
  - Randwick
  - Richmond
- Austria (7):
  - Feldkirch
  - Gratwein
  - Graz
  - Hartberg
  - Linz
  - Vienna
  - Zams
- Belgium (5):
  - Brussels
  - Huy
  - Leper
  - Leuven
  - Yvoir
- Brazil (13):
  - Belo Horizonte - MG
  - Botucatu
  - Brasilia/DF
  - Brasília
  - Campinas
  - Campinas, Sao Paulo
  - Curitiba - PR
  - Porto Alegre
  - Porto Alegre/RS
  - Salvador
  - Salvador/BA
  - São José Do Rio Preto- SP
  - São Paulo
- Bulgaria (7):
  - Gabrovo
  - Pleven
  - Plovdiv
  - Sandanski
  - Sliven
  - Sofia
  - Yambol
- Canada (9):
  - Edmonton, Alberta
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Kitchener, Ontario
  - Ottawa, Ontario
  - Thunder Bay, Ontario
  - Montreal, Quebec
  - Ontario
  - Québec
- Chile (5):
  - La Serena
  - Osorno
  - Santiago
  - Temuco
  - Viña del Mar
- Croatia (6):
  - Krapinske Toplice
  - Pula
  - Rijeka
  - Varaždin
  - Zadar
  - Zagreb
- Czechia (18):
  - Chrudim
  - Čáslav
  - Hradec Králové
  - Kladno
  - Kroměříž
  - Kyjov
  - Liberec
  - Litomyšl
  - Olomouc
  - Ostrava
  - Plzen - Bory
  - Prague
  - Slaný
  - Strakonice
  - Teplice
  - Ústí nad Labem
  - Zlín
  - Znojmo
- Denmark (10):
  - Aarhus N
  - Frederiksberg
  - Glostrup Municipality
  - Haderslev
  - Hellerup
  - Hillerød
  - Hvidovre
  - København NV
  - Silkeborg
  - Slagelse
- Estonia (2):
  - Tallinn
  - Tartu
- Finland (7):
  - Helsinki
  - Jyväskylä
  - Kouvola
  - Mikkeli
  - Pori
  - Tampere
  - Turku
- France (26):
  - Angers
  - Arras
  - Avignon
  - Bois-Guillaume
  - Bordeaux
  - Brest
  - Cambrai
  - Castelnau-le-Lez
  - Clermont-Ferrand
  - Colombes
  - Dijon
  - La Tronche
  - Le Mans
  - Lille
  - Limoges
  - Montpellier
  - Nantes
  - Nîmes
  - Paris
  - Pierre-Bénite
  - Quimper
  - Rennes
  - Saint-Priest En Jarrez
  - Tourcoing
  - Valenciennes
  - Vernon
- Tbilisi, Georgia
- Germany (23):
  - Altenburg
  - Bad Friedrichshall
  - Berlin
  - Bonn
  - Dresden
  - Essen
  - Hamburg
  - Heidelberg
  - Karlbad
  - Ludwigshafen
  - Magdeburg
  - Mainz
  - Minden
  - Möchengladbach
  - Neuss
  - Oberhausen
  - Paderborn
  - Rüsselsheim am Main
  - Troisdorf
  - Weiden
  - Wesel
  - Wiesbaden
  - Witten
- Hungary (17):
  - Baja
  - Balassagyarmat
  - Balatonfüred
  - Berettyóújfalu
  - Budapest
  - Cegléd
  - Debrecen
  - Eger
  - Gyula
  - Hódmezövásárhely
  - Kistarcsa
  - Mohács
  - Nagykanizsa
  - Szekszárd
  - Szolnok
  - Veszprém
  - Zalaegerszeg
- Israel (9):
  - Afula
  - Ashkelon
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Safed
  - Tel Aviv
  - Ẕerifin
- Italy (14):
  - Castelfranco Veneto, Treviso
  - Bollate
  - Frenze
  - Genova
  - Milan
  - Napoli
  - Parma
  - Pavia
  - Piacenza
  - Reggio Emilia
  - Roma
  - Varese
  - Venezia
  - Vittorio Veneto TV
- Latvia (4):
  - Daugavpils
  - Liepāja
  - Riga
  - Valmiera
- Lithuania (6):
  - Alytus
  - Kaunas
  - Klaipėda
  - Šiauliai
  - Utena
  - Vilnius
- Picayune, MS, Montserrat
- Peru (3):
  - Arequipa
  - Callao
  - Lima
- Poland (9):
  - Bialystok
  - Bydgoszcz
  - Czeladź
  - Gdansk
  - Krakow
  - Skierniewice
  - Tarnobrzeg
  - Warsaw
  - Włocławek
- Romania (9):
  - Baia
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Iași
  - Oradea
  - Piteşti
  - Târgu Mureş
  - Timișoara
- Russia (22):
  - Arkhangelsk
  - Barnaul
  - Belgorod
  - Chelyabinsk
  - Irkutsk
  - Kaluga
  - Kazan'
  - Kemerovo
  - Kirov
  - Krasnodar
  - Lubertsy
  - Moscow
  - Murmansk
  - Novosibirsk
  - Rostov-on-Don
  - Saint Petersburg
  - Samara
  - Saratov
  - Smolensk
  - Tomsk
  - Yaroslavl
  - Yekaterinburg
- Serbia (6):
  - Belgrade
  - Kamenitz
  - Kragujevac
  - Niš
  - Niška Banja
  - Pančevo
- Singapore, Singapore
- Slovakia (2):
  - Bratislava
  - Nitra
- South Africa (4):
  - Johannesburg, Gauteng
  - Cape Town, Western Cape
  - Pretoria
  - Worcester
- Spain (18):
  - Barcelona, Catalonia
  - L'Hospitalet de Llobregat, Catalonia
  - Sabadell, Catalonia
  - Sant Boi de Llobregat, Catalonia
  - Tarragona, Catalonia
  - Madrid, Communidad de
  - Vigo, Galicia
  - Madrid, Madrid, Communidad de
  - Majadahonda, Madrid, Communidad de
  - San Sebastián de los Reyes, Madrid, Communidad de
  - Orihuela, Valencia
  - Barcelona
  - Cartagena
  - Girona
  - Olot
  - Pontevedra
  - Salamanca
  - Terrassa
- Ukraine (16):
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kherson
  - Kirovograd
  - Kyiv
  - Luhansk
  - Lutsk
  - Lviv
  - Odesa
  - Rivne
  - Simferopol
  - Uzhhorod
  - Vinnytsia
  - Yevpatoria
  - Zaporizhzhya
- United Kingdom (5):
  - London
  - Manchester
  - Newcastle upon Tyne
  - Romford
  - Southall

REFERENCES:
- [Derived] Chi G, Violi F, Pignatelli P, Vestri A, Spagnoli A, Loffredo L, Hernandez AF, Hull RD, Cohen AT, Harrington RA, Goldhaber SZ, Gibson CM. External validation of the ADA score for predicting thrombosis among acutely ill hospitalized medical patients from the APEX Trial. J Thromb Thrombolysis. 2023 Feb;55(2):211-221. doi: 10.1007/s11239-022-02757-8. Epub 2022 Dec 24. PMID 36566304
- [Derived] Jamil A, Jamil U, Singh K, Khan F, Chi G. Extended Thromboprophylaxis With Betrixaban or Rivaroxaban for Acutely Ill Hospitalized Medical Patients: Meta-Analysis of Prespecified Subgroups. Crit Pathw Cardiol. 2021 Mar 1;20(1):16-24. doi: 10.1097/HPC.0000000000000232. PMID 32657973
- [Derived] Yee MK, Gibson CM, Nafee T, Kerneis M, Daaboul Y, Korjian S, Chi G, AlKhalfan F, Hernandez AF, Hull RD, Cohen AT, Goldhaber SZ. Characterization of Major and Clinically Relevant Non-Major Bleeds in the APEX Trial. TH Open. 2019 Apr 17;3(2):e103-e108. doi: 10.1055/s-0039-1685496. eCollection 2019 Apr. PMID 31249989
- [Derived] Guy H, Laskier V, Fisher M, Bucior I, Deitelzweig S, Cohen AT. Budget impact analysis of betrixaban for venous thromboembolism prophylaxis in nonsurgical patients with acute medical illness in the United Kingdom. Expert Rev Pharmacoecon Outcomes Res. 2020 Jun;20(3):259-267. doi: 10.1080/14737167.2019.1629905. Epub 2019 Jun 19. PMID 31215264
- [Derived] Chi G, Gibson CM, Kalayci A, Cohen AT, Hernandez AF, Hull RD, Kahe F, Jafarizade M, Sharfaei S, Liu Y, Harrington RA, Goldhaber SZ. Extended-duration betrixaban versus shorter-duration enoxaparin for venous thromboembolism prophylaxis in critically ill medical patients: an APEX trial substudy. Intensive Care Med. 2019 Apr;45(4):477-487. doi: 10.1007/s00134-019-05565-6. Epub 2019 Feb 18. PMID 30778649
- [Derived] Kalayci A, Gibson CM, Chi G, Yee MK, Korjian S, Datta S, Nafee T, Gurin M, Haroian N, Qamar I, Hull RD, Hernandez AF, Cohen AT, Harrington RA, Goldhaber SZ. Asymptomatic Deep Vein Thrombosis is Associated with an Increased Risk of Death: Insights from the APEX Trial. Thromb Haemost. 2018 Dec;118(12):2046-2052. doi: 10.1055/s-0038-1675606. Epub 2018 Nov 12. PMID 30419597
- [Derived] Chi G, Gibson CM, Liu Y, Hernandez AF, Hull RD, Cohen AT, Harrington RA, Goldhaber SZ. Inverse relationship of serum albumin to the risk of venous thromboembolism among acutely ill hospitalized patients: Analysis from the APEX trial. Am J Hematol. 2019 Jan;94(1):21-28. doi: 10.1002/ajh.25296. Epub 2018 Oct 17. PMID 30252149
- [Derived] Chi G, Goldhaber SZ, Hull RD, Hernandez AF, Kerneis M, Al Khalfan F, Cohen AT, Harrington RA, Gibson CM. Thrombus Burden of Deep Vein Thrombosis and Its Association with Thromboprophylaxis and D-Dimer Measurement: Insights from the APEX Trial. Thromb Haemost. 2017 Dec;117(12):2389-2395. doi: 10.1160/TH17-08-0538. Epub 2017 Dec 6. PMID 29212126
- [Derived] Yee MK, Nafee T, Daaboul Y, Korjian S, AlKhalfan F, Kerneis M, Wiest C, Goldhaber SZ, Hernandez AF, Hull RD, Cohen AT, Harrington RA, Gibson CM. Increased benefit of betrixaban among patients with a history of venous thromboembolism: a post-hoc analysis of the APEX trial. J Thromb Thrombolysis. 2018 Jan;45(1):1-8. doi: 10.1007/s11239-017-1583-0. PMID 29188425
- [Derived] Chi G, Januzzi JL, Korjian S, Daaboul Y, Goldhaber SZ, Hernandez AF, Hull RD, Gold A, Cohen AT, Harrington RA, Gibson CM. N-terminal pro-B-type natriuretic peptide and the risk of stroke among patients hospitalized with acute heart failure: an APEX trial substudy. J Thromb Thrombolysis. 2017 Nov;44(4):457-465. doi: 10.1007/s11239-017-1552-7. PMID 28905172
- [Derived] Arbetter DF, Jain P, Yee MK, Michalak N, Hernandez AF, Hull RD, Goldhaber SZ, Harrington RA, Gold A, Cohen AT, Gibson CM. Competing risk analysis in a large cardiovascular clinical trial: An APEX substudy. Pharm Stat. 2017 Nov;16(6):445-450. doi: 10.1002/pst.1823. Epub 2017 Aug 24. PMID 28840662
- [Derived] Chi G, Goldhaber SZ, Kittelson JM, Turpie AGG, Hernandez AF, Hull RD, Gold A, Curnutte JT, Cohen AT, Harrington RA, Gibson CM. Effect of extended-duration thromboprophylaxis on venous thromboembolism and major bleeding among acutely ill hospitalized medical patients: a bivariate analysis. J Thromb Haemost. 2017 Oct;15(10):1913-1922. doi: 10.1111/jth.13783. Epub 2017 Sep 4. PMID 28762617
- [Derived] Gibson CM, Korjian S, Chi G, Daaboul Y, Jain P, Arbetter D, Goldhaber SZ, Hull R, Hernandez AF, Lopes RD, Gold A, Cohen AT, Harrington RA; APEX Investigators. Comparison of Fatal or Irreversible Events With Extended-Duration Betrixaban Versus Standard Dose Enoxaparin in Acutely Ill Medical Patients: An APEX Trial Substudy. J Am Heart Assoc. 2017 Jul 11;6(7):e006015. doi: 10.1161/JAHA.117.006015. PMID 28698258
- [Derived] Gibson CM, Goldhaber SZ, Cohen AT, Nafee T, Hernandez AF, Hull R, Korjian S, Daaboul Y, Chi G, Yee M, Harrington RA. When academic research organizations and clinical research organizations disagree: Processes to minimize discrepancies prior to unblinding of randomized trials. Am Heart J. 2017 Jul;189:1-8. doi: 10.1016/j.ahj.2017.03.018. Epub 2017 Mar 31. No abstract available. PMID 28625365
- [Derived] Marszalek J, Mehrsefat S, Chi G. The risk of stroke among acutely ill hospitalized medical patients: lessons from recent trials on extended-duration thromboprophylaxis. Expert Rev Hematol. 2017 Aug;10(8):679-684. doi: 10.1080/17474086.2017.1343662. Epub 2017 Jun 21. PMID 28617144
- [Derived] Gibson CM, Chi G, Halaby R, Korjian S, Daaboul Y, Jain P, Arbetter D, Goldhaber SZ, Hull R, Hernandez AF, Gold A, Bandman O, Harrington RA, Cohen AT; APEX Investigators. Extended-Duration Betrixaban Reduces the Risk of Stroke Versus Standard-Dose Enoxaparin Among Hospitalized Medically Ill Patients: An APEX Trial Substudy (Acute Medically Ill Venous Thromboembolism Prevention With Extended Duration Betrixaban). Circulation. 2017 Feb 14;135(7):648-655. doi: 10.1161/CIRCULATIONAHA.116.025427. Epub 2016 Nov 14. PMID 27881569
- [Derived] Cohen AT, Harrington RA, Goldhaber SZ, Hull RD, Wiens BL, Gold A, Hernandez AF, Gibson CM; APEX Investigators. Extended Thromboprophylaxis with Betrixaban in Acutely Ill Medical Patients. N Engl J Med. 2016 Aug 11;375(6):534-44. doi: 10.1056/NEJMoa1601747. Epub 2016 May 27. PMID 27232649
- [Derived] Cohen AT, Harrington R, Goldhaber SZ, Hull R, Gibson CM, Hernandez AF, Kitt MM, Lorenz TJ. The design and rationale for the Acute Medically Ill Venous Thromboembolism Prevention with Extended Duration Betrixaban (APEX) study. Am Heart J. 2014 Mar;167(3):335-41. doi: 10.1016/j.ahj.2013.11.006. Epub 2013 Dec 10. PMID 24576517

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was enrolled on 3/29/2012 and last patient completed the study on 1/15/2016. Patients meeting the inclusion and none of the exclusion criteria at screening were randomized 1:1 to either the betrixaban or enoxaparin treatment group.
Pre-assignment Details: To maintain the blind, patients either received betrixaban capsules for 35 to 42 days and daily subcutaneous (SQ) injections of enoxaparin placebo for 10 ± 4 days, or received daily SQ injections of enoxaparin for 10 ± 4 days and betrixaban placebo capsules for 35 to 42 days.
Period: Overall Study
Arm/Group | Betrixaban | Enoxaparin
Started | 3759 | 3754
Completed | 3470 | 3471
Not Completed | 289 | 283
Not completed — Withdrawal by Subject | 43 | 29
Not completed — Death | 206 | 211
Not completed — Lost to Follow-up | 11 | 17
Not completed — Adverse event or serious adverse event | 3 | 3
Not completed — Patient /Family decision | 3 | 0
Not completed — Cannot contact patient directly | 1 | 2
Not completed — SOURCE DOCUMENT/COORDINATOR MISSING | 0 | 2
Not completed — Patient did not wish to attend visits | 0 | 1
Not completed — Patient randomized but not dosed | 17 | 16
Not completed — Patient was assessed via phone in person | 1 | 0
Not completed — Patient deemed ineligible after random | 2 | 0
Not completed — Patient was early terminated from study | 0 | 1
Not completed — Patient was randomized due to mistake | 1 | 0
Not completed — THE SUBJECT MOVED TO ANOTHER PROVINCE | 0 | 1
Not completed — Withdraw of consent on day of random | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Betrixaban | Enoxaparin | Total
Number analyzed (Participants) | 3759 | 3754 | 7513
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.6 (8.46) | 76.2 (8.31) | 76.4 (8.39)
Age, Customized [Count of Participants; unit: Participants]
  <75 years | 1184 | 1237 | 2421
  >=75 years | 2575 | 2517 | 5092
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2054 | 2034 | 4088
  Male | 1705 | 1720 | 3425

OUTCOME MEASURES:

1. Primary Outcome: Modified Intent-to-Treat (mITT) Cohort 1: Percentage of Participants Experiencing the Composite Event of Symptomatic Deep Vein Thrombosis (DVT), Non-fatal Pulmonary Emboli (PE), VTE-related Death, or Asymptomatic Proximal DVT, Through Visit 3
Description: mITT Cohort 1: Percentage of participants experiencing either symptomatic DVT, non-fatal PE, venous thromboembolism (VTE) related death adjudicated by a blinded independent Clinical Events Committee (CEC) between randomization and on or before Visit 3 or Day 42 if patient did not have a Visit 3, or a blinded ultrasound core laboratory measuring of asymptomatic proximal DVT between randomization and Day 47. Visit 3 is between day 35-42 after randomization (day 1).
Time Frame: mITT Cohort 1: Between randomization and Day 47 (max)
Population: Cohort 1 (participants with baseline D-dimer ≥ 2 x upper limit normal (ULN) as determined by the local lab) of the mITT population which consisted of all participants who had taken at least one dose of study drug and who had follow-up assessment data on one or more primary or secondary efficacy components.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Betrixaban | Enoxaparin
Number analyzed (Participants) | 2314 | 2313
Percentage of Participants | 5.70 [4.76 to 6.65] | 7.18 [6.12 to 8.23]
Statistical Analysis 1: Comparison: Betrixaban vs Enoxaparin; Test type: Superiority; p = 0.038, Cochran-Mantel-Haenszel; Relative Risk Reduction (RRR) = 0.209, 95% CI 2-sided [0.013 to 0.366]

2. Primary Outcome: mITT Cohort 2: Percentage of Participants Experiencing the Composite Event of Symptomatic DVT, Non-fatal PE, VTE-related Death, or Asymptomatic Proximal DVT, Through Visit 3
Description: mITT Cohort 2: Percentage of participants experiencing either symptomatic DVT, non-fatal PE, VTE related death adjudicated by a blinded independent CEC between randomization and on or before Visit 3 or Day 42 if patient did not have a Visit 3, or a blinded ultrasound core laboratory measuring of asymptomatic proximal DVT between randomization and Day 47. Visit 3 is between day 35-42 after randomization (day 1).
Time Frame: mITT Cohort 2: Between randomization and Day 47 (max)
Population: Cohort 2 (encompasses "both" participants over 75 and participants with baseline D-dimer ≥ 2 x ULN as determined by the local lab) of the mITT population which consisted of all participants who had taken at least one dose of study drug and who had follow-up assessment data on one or more primary or secondary efficacy components.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Betrixaban | Enoxaparin
Number analyzed (Participants) | 3407 | 3391
Percentage of Participants | 4.70 [3.99 to 5.41] | 6.02 [5.22 to 6.82]
Statistical Analysis 1: Comparison: Betrixaban vs Enoxaparin; Test type: Superiority; p = 0.018, Cochran-Mantel-Haenszel; Relative Risk Reduction (RRR) = 0.216, 95% CI 2-sided [0.041 to 0.359]

3. Primary Outcome: mITT: Percentage of Participants Experiencing the Composite Event of Symptomatic DVT, Non-fatal PE, VTE-related Death, or Asymptomatic Proximal DVT, Through Visit 3
Description: mITT: Percentage of participants experiencing either symptomatic DVT, non-fatal PE, VTE related death adjudicated by a blinded independent CEC between randomization and on or before Visit 3 or Day 42 if patient did not have a Visit 3, or a blinded ultrasound core laboratory measuring of asymptomatic proximal DVT between randomization and Day 47. Visit 3 is between day 35-42 after randomization (day 1).
Time Frame: mITT: Between randomization and Day 47 (max)
Population: The mITT population which consisted of all participants who had taken at least one dose of study drug and who had follow-up assessment data on one or more primary or secondary efficacy components.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Betrixaban | Enoxaparin
Number analyzed (Participants) | 3721 | 3720
Percentage of Participants | 4.43 [3.77 to 5.10] | 5.99 [5.23 to 6.76]
Statistical Analysis 1: Comparison: Betrixaban vs Enoxaparin; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Relative Risk Reduction (RRR) = 0.254, 95% CI 2-sided [0.092 to 0.387]

4. Primary Outcome: Percentage of Participants Experiencing Major Bleeding Through Seven Days After Discontinuation of All Study Medication
Description: Percentage of participants experiencing at least one major bleeding adjudicated by a blinded independent CEC between randomization (day 1) and up to seven days after discontinuation of all study medication.
Time Frame: Between randomization and Day 49 (max)
Population: Safety population which consisted of all participants who had taken at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Betrixaban | Enoxaparin
Number analyzed (Participants) | 3716 | 3716
Percentage of Participants | 0.67 [0.41 to 0.94] | 0.57 [0.32 to 0.81]
Statistical Analysis 1: Comparison: Betrixaban vs Enoxaparin; Test type: Superiority; p = 0.554, Chi-squared

5. Secondary Outcome: mITT Cohort 1: Percentage of Participants Experiencing the Composite Event of Symptomatic DVT, Non-fatal PE, or VTE-related Death, Through Visit 3
Description: mITT Cohort 1: Percentage of participants experiencing either symptomatic DVT, non-fatal PE, or VTE related death adjudicated by a blinded independent CEC between randomization and on or before Visit 3 or Day 42 if patient did not have a Visit 3. Visit 3 is between day 35-42 after randomization (day 1).
Time Frame: mITT Cohort 1: Between randomization and Day 42 (max)
Population: Cohort 1 (participants with baseline D-dimer ≥ 2 x ULN as determined by the local lab) of the mITT population which consisted of all participants who had taken at least one dose of study drug and who had follow-up assessment data on one or more primary or secondary efficacy components.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Betrixaban | Enoxaparin
Number analyzed (Participants) | 2314 | 2313
Percentage of Participants | 1.30 [0.84 to 1.76] | 1.90 [1.35 to 2.46]
Statistical Analysis 1: Comparison: Betrixaban vs Enoxaparin; Test type: Superiority; p = 0.092, Cochran-Mantel-Haenszel; Relative Risk Reduction (RRR) = 0.326, 95% CI 2-sided [-0.069 to 0.576]

6. Secondary Outcome: mITT Cohort 2: Percentage of Participants Experiencing the Composite Event of Symptomatic DVT, Non-fatal PE, or VTE-related Death, Through Visit 3
Description: mITT Cohort 2: Percentage of participants experiencing either symptomatic DVT, non-fatal PE, or VTE related death adjudicated by a blinded independent CEC between randomization and on or before Visit 3 or Day 42 if patient did not have a Visit 3. Visit 3 is between day 35-42 after randomization (day 1).
Time Frame: mITT Cohort 2: Between randomization and Day 42 (max)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Betrixaban | Enoxaparin
Number analyzed (Participants) | 3407 | 3391
Percentage of Participants | 1.03 [0.69 to 1.37] | 1.45 [1.04 to 1.85]
Statistical Analysis 1: Comparison: Betrixaban vs Enoxaparin; Test type: Superiority; p = 0.11, Cochran-Mantel-Haenszel; Relative Risk Reduction (RRR) = 0.295, 95% CI 2-sided [-0.085 to 0.542]

7. Secondary Outcome: mITT: Percentage of Participants Experiencing the Composite Event of Symptomatic DVT, Non-fatal PE, or VTE-related Death, Through Visit 3
Description: mITT: Percentage of participants experiencing either symptomatic DVT, non-fatal PE, or VTE related death adjudicated by a blinded independent CEC between randomization and on or before Visit 3 or Day 42 if patient did not have a Visit 3. Visit 3 is between day 35-42 after randomization (day 1).
Time Frame: mITT: Between randomization and Day 42 (max)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Betrixaban | Enoxaparin
Number analyzed (Participants) | 3721 | 3720
Percentage of Participants | 0.94 [0.63 to 1.25] | 1.45 [1.07 to 1.84]
Statistical Analysis 1: Comparison: Betrixaban vs Enoxaparin; Test type: Superiority; p = 0.039, Cochran-Mantel-Haenszel; Relative Risk Reduction (RRR) = 0.358, 95% CI 2-sided [0.020 to 0.580]

ADVERSE EVENTS:
Time Frame: From first dose date (including) till the end of study
Description: The number of patients at risk by study arm in the Adverse Events Results is based on Safety population, defined as patients who were randomized and received at least one dose of study drug. It leads to 3716 safety subjects in Betrixaban arm and 3716 in Enoxaprin arm which corresponds to the number of patients at risk in Adverse Events Results.
Arm/Group | Betrixaban | Enoxaparin
Serious Adverse Events (participants affected / at risk) | 657/3716 | 615/3716
Other Adverse Events (participants affected / at risk) | 879/3716 | 779/3716
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Betrixaban (N=3716) | Enoxaparin (N=3716)
Cardiac failure (Cardiac disorders) | 83 | 66
Atrial fibrillation (Cardiac disorders) | 11 | 23
Cardiac failure congestive (Cardiac disorders) | 10 | 15
Cardiac failure acute (Cardiac disorders) | 10 | 12
Cardiac failure chronic (Cardiac disorders) | 13 | 9
Acute myocardial infarction (Cardiac disorders) | 6 | 12
Myocardial infarction (Cardiac disorders) | 7 | 10
Cardiogenic shock (Cardiac disorders) | 9 | 6
Cardiac arrest (Cardiac disorders) | 7 | 5
Coronary artery disease (Cardiac disorders) | 8 | 3
Angina unstable (Cardiac disorders) | 3 | 7
Acute coronary syndrome (Cardiac disorders) | 6 | 3
Atrioventricular block complete (Cardiac disorders) | 5 | 3
Myocardial ischaemia (Cardiac disorders) | 2 | 6
Angina pectoris (Cardiac disorders) | 5 | 0
Cardio-respiratory arrest (Cardiac disorders) | 3 | 2
Cardiopulmonary failure (Cardiac disorders) | 1 | 4
Ventricular tachycardia (Cardiac disorders) | 4 | 1
Coronary artery insufficiency (Cardiac disorders) | 2 | 2
Atrioventricular block (Cardiac disorders) | 1 | 2
Cardiovascular disorder (Cardiac disorders) | 1 | 2
Cardiovascular insufficiency (Cardiac disorders) | 0 | 3
Ventricular fibrillation (Cardiac disorders) | 1 | 2
Atrial flutter (Cardiac disorders) | 0 | 2
Atrioventricular block second degree (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 2 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 1
Cor pulmonale (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Pericardial haemorrhage (Cardiac disorders) | 1 | 0
Sinoatrial block (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0
Trifascicular block (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular hypokinesia (Cardiac disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 38 | 43
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 30 | 17
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 | 26
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 46 | 64
Urinary tract infection (Infections and infestations) | 13 | 11
Sepsis (Infections and infestations) | 13 | 7
Septic shock (Infections and infestations) | 7 | 8
Cellulitis (Infections and infestations) | 3 | 7
Bronchitis (Infections and infestations) | 1 | 6
Respiratory tract infection (Infections and infestations) | 4 | 3
Erysipelas (Infections and infestations) | 4 | 2
Gastroenteritis (Infections and infestations) | 4 | 0
Bronchopneumonia (Infections and infestations) | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 2
Endocarditis (Infections and infestations) | 1 | 2
Infected skin ulcer (Infections and infestations) | 2 | 1
Lobar pneumonia (Infections and infestations) | 1 | 2
Pyelonephritis (Infections and infestations) | 2 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 2
Wound infection (Infections and infestations) | 2 | 1
Appendicitis (Infections and infestations) | 1 | 1
Clostridium colitis (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 2 | 0
Pseudomembranous colitis (Infections and infestations) | 2 | 0
Pulmonary sepsis (Infections and infestations) | 2 | 0
Pulmonary tuberculosis (Infections and infestations) | 2 | 0
Tracheobronchitis (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 1
Abscess bacterial (Infections and infestations) | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bone abscess (Infections and infestations) | 1 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 1 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0
Gallbladder empyema (Infections and infestations) | 0 | 1
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 1 | 0
Nosocomial infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Psoas abscess (Infections and infestations) | 1 | 0
Pyelocystitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 19 | 35
Brain oedema (Nervous system disorders) | 8 | 10
Cerebrovascular accident (Nervous system disorders) | 7 | 6
Syncope (Nervous system disorders) | 4 | 4
Cerebral infarction (Nervous system disorders) | 3 | 3
Transient ischaemic attack (Nervous system disorders) | 2 | 4
Convulsion (Nervous system disorders) | 2 | 3
Loss of consciousness (Nervous system disorders) | 4 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 2
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 2
Coma (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 2
Epilepsy (Nervous system disorders) | 1 | 1
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 1 | 0
Neuroglycopenia (Nervous system disorders) | 1 | 0
Neurological decompensation (Nervous system disorders) | 0 | 1
Paralysis flaccid (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 18 | 5
Rectal haemorrhage (Gastrointestinal disorders) | 15 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 3 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 4
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 4
Colitis (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 0
Melaena (Gastrointestinal disorders) | 1 | 1
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 16 | 38
Hypotension (Vascular disorders) | 8 | 3
Haematoma (Vascular disorders) | 5 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 2
Peripheral ischaemia (Vascular disorders) | 1 | 2
Aortic aneurysm (Vascular disorders) | 1 | 1
Aortic dissection (Vascular disorders) | 1 | 1
Aortic stenosis (Vascular disorders) | 2 | 0
Arteriosclerosis (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 2 | 0
Haemorrhagic vasculitis (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1
Venous thrombosis (Vascular disorders) | 0 | 2
Aneurysm (Vascular disorders) | 0 | 1
Angiopathy (Vascular disorders) | 1 | 0
Arterial disorder (Vascular disorders) | 1 | 0
Arterial stenosis (Vascular disorders) | 1 | 0
Bleeding varicose vein (Vascular disorders) | 1 | 0
Embolism arterial (Vascular disorders) | 1 | 0
Essential hypertension (Vascular disorders) | 1 | 0
Femoral artery aneurysm (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Intra-abdominal haematoma (Vascular disorders) | 0 | 1
Ischaemia (Vascular disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Phlebitis superficial (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 10 | 15
Renal failure acute (Renal and urinary disorders) | 12 | 11
Haematuria (Renal and urinary disorders) | 17 | 5
Renal failure chronic (Renal and urinary disorders) | 8 | 4
Haemorrhage urinary tract (Renal and urinary disorders) | 2 | 1
Renal impairment (Renal and urinary disorders) | 3 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0
Death (General disorders) | 9 | 16
Sudden cardiac death (General disorders) | 6 | 5
Multi-organ failure (General disorders) | 3 | 6
General physical health deterioration (General disorders) | 6 | 2
Sudden death (General disorders) | 3 | 3
Non-cardiac chest pain (General disorders) | 2 | 1
Pyrexia (General disorders) | 3 | 0
Cardiac death (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 1
Condition aggravated (General disorders) | 1 | 0
Device malfunction (General disorders) | 1 | 0
Discomfort (General disorders) | 0 | 1
Fibrosis (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 1
Hyperthermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 1
Necrosis (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Puncture site haemorrhage (General disorders) | 0 | 1
Ulcer (General disorders) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 8
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 3
Fall (Injury, poisoning and procedural complications) | 3 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 3
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Iatrogenic injury (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 8 | 4
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0
Hepatic enzyme increased (Investigations) | 2 | 5
Aspiration bronchial (Investigations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
General physical condition abnormal (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Blood urine present (Investigations) | 1 | 0
Catheterisation cardiac (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 4 | 0
Bile duct stone (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 2 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Coronary artery bypass (Surgical and medical procedures) | 1 | 0
Glaucoma surgery (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0
Hysterectomy (Surgical and medical procedures) | 1 | 0
Leg amputation (Surgical and medical procedures) | 0 | 1
Mitral valve repair (Surgical and medical procedures) | 0 | 1
Surgery (Surgical and medical procedures) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Goitre (Endocrine disorders) | 1 | 0
Hypoparathyroidism (Endocrine disorders) | 0 | 1
Activities of daily living impaired (Social circumstances) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Betrixaban (N=3716) | Enoxaparin (N=3716)
Urinary tract infection (Infections and infestations) | 110 | 78
Constipation (Gastrointestinal disorders) | 109 | 102
Hypokalaemia (Metabolism and nutrition disorders) | 91 | 84
Hypertension (Vascular disorders) | 88 | 80
Insomnia (Psychiatric disorders) | 87 | 89
Headache (Nervous system disorders) | 74 | 59
Nausea (Gastrointestinal disorders) | 67 | 55
Diarrhoea (Gastrointestinal disorders) | 63 | 59
Renal cyst (Renal and urinary disorders) | 55 | 47
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 53 | 41
Atrial fibrillation (Cardiac disorders) | 50 | 85
Cardiac failure (Cardiac disorders) | 48 | 32
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 48 | 19
Haematuria (Renal and urinary disorders) | 46 | 23
Anaemia (Blood and lymphatic system disorders) | 44 | 29
Mitral valve incompetence (Cardiac disorders) | 41 | 49
Oedema peripheral (General disorders) | 39 | 19
Tricuspid valve incompetence (Cardiac disorders) | 38 | 41
Deep vein thrombosis (Vascular disorders) | 29 | 58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Due to multi centers, studies and countries this varies.